CLINICAL TRIAL: NCT01214005
Title: Smoking Abstinence and Lapse Effects in Smokers With Schizophrenia and Controls
Acronym: WREN
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brown University (Other)
Responsible Party: Principal Investigator, Jennifer Tidey, Associate Professor (Research), Brown University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: R21DA026829 (NIH)
Record Dates: First submitted 2010-10-01; First posted 2010-10-04 (Estimated); Last update posted 2012-04-27 (Estimated); Status verified 2012-04

CONDITIONS: Tobacco Use Disorder; Schizophrenia
Keywords: nicotine; reinforcement; craving; relapse
MeSH Terms: conditions — Tobacco Use Disorder; Schizophrenia; Recurrence

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- schizophrenia (Experimental): Smokers with schizophrenia or schizoaffective disorder
  Interventions: Behavioral: smoking abstinence
- non-psychiatric (Other): smokers without psychiatric illness
  Interventions: Behavioral: smoking abstinence

INTERVENTIONS:
Behavioral: smoking abstinence — 3 days of biologically-confirmed smoking abstinence

SUMMARY:
This project tests two hypotheses concerning the low smoking cessation rates in smokers with schizophrenia. The first hypothesis is that smokers with schizophrenia experience stronger and more sustained effects of smoking abstinence on negative mood and smoking urge than control smokers without psychiatric illness. The second hypothesis is that smokers with schizophrenia experience stronger reinforcing effects of a smoking lapse (i.e., more rewarding effects of smoking after a period of abstinence) than control smokers without psychiatric illness.

DETAILED DESCRIPTION:
In this study, smokers with schizophrenia and smokers without psychiatric illness participate in a nicotine preference task before and after a 3-day period of continuous smoking abstinence. The investigators will experimentally control abstinence by providing participants with high-value cash incentives contingent upon smoking abstinence verified with breath carbon monoxide levels. The investigators will measure nicotine withdrawal and smoking urge during the abstinence period. In the nicotine preference task, participants will make choices between nicotine-containing and denicotinized cigarette puffs to provide a measure of nicotine reinforcement, and the investigators will also measure the effects of smoking on mood. After the second nicotine preference task, participants will receive a small-value reinforcer if they continue to abstain for another day, and the investigators will measure time to the second lapse.

ELIGIBILITY:
Inclusion Criteria:

* cigarette smokers, 20-50 cigarettes per day
* schizophrenia or no psychiatric illness
* age 18 or older
* male or female

Exclusion Criteria:

* unstable symptoms or medication
* not interested in quitting smoking within 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Withdrawal symptoms | 3 days
  negative mood related to nicotine withdrawal
urge to smoke | 3 days
  craving for smoking
nicotine preference | before and after 3 days of abstinence
  choice for nicotine puffs versus denicotinized cigarette puffs
positive and negative mood | before and after 3 days of abstinence
  positive and negative mood scale

SECONDARY OUTCOMES:
time to lapse | 192 hours
  time between smoking behavior in the laboratory and first cigarette outside of the laboratory

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Tidey, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, 121 South Main Street, Providence, Rhode Island, United States